CLINICAL TRIAL: NCT00221351
Title: A Randomized, Controlled Trial of a C-reactive Protein (CRP)-Guided Management Algorithm for Adults With Acute Cough Illness in the Emergency Department
Brief Title: C-reactive Protein (CRP)-Guided Management Algorithm for Adults With Acute Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRP-1; IMPAACT- AHRQ/ VAMC
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Cough
Keywords: cough; acute bronchitis; upper respiratory tract infection; pneumonia; lower respiratory tract infection
MeSH Terms: conditions — Cough; Bronchitis; Respiratory Tract Infections; Pneumonia

INTERVENTIONS:
Procedure: CRP point of care testing

SUMMARY:
We aim to evaluate the impact of a CRP-guided management algorithm for adults with acute cough illness. More specifically, we will examine both process of care and clinical outcomes:

1. Processes of care (i.e., chest x-rays ordered, antibiotic treatment, length-of-time in the ED). We hypothesize that CRP-guided management will be associated with a decrease in the antibiotic prescription for acute cough illness from 50 percent to 30 percent.
2. Clinical outcomes (i.e., duration of illness, any return visit, return visit with a diagnosis of pneumonia, hospitalization, subsequent antibiotic use, satisfaction with care). We hypothesize that there will be no difference in the proportion of patients feeling back to normal within 2 weeks of their ED visit for acute cough illness (about 60 percent, 95% confidence interval=50 to 70 percent).

DETAILED DESCRIPTION:
We have developed a CRP-guided management algorithm based on recent studies in which the accuracy of CRP for identifying patients with pneumonia was confirmed.(10;11) Importantly, these 2 studies each confirmed that CRP levels provide additional diagnostic support beyond that gained from application of clinical prediction rules. In the proposed study, we will recommend that physicians first assess the probability of pneumonia based on clinical findings, in accordance with current practice recommendations as follows: 1) Low Clinical Suspicion (<5% probability of pneumonia): Absence of fever (T>38C), tachycardia (HR>100), or tachypnea (RR>24), and normal chest examination. These patients should receive symptomatic therapy, and do not require CXR or antibiotic treatment; 2) High Clinical Suspicion (>30% probability of pneumonia): At least 1 abnormal vital sign and abnormal chest examination. These patients receive CXR and antibiotics based on CXR findings or high clinical suspicion; 3) Intermediate Clinical Suspicion (5-30%): All others. Current practice guidelines recommend considering CXR in these patients, however no further guidance is provided for the management of these patients.

After assessing the clinical probability of pneumonia, CRP levels will be provided for a random subset of patients. A CRP level <10 mg/L corresponds with a very low probability of bacterial pneumonia. Thus, for patients with low and intermediate-probability of pneumonia based on clinical grounds, a CRP <10 mg/L should confirm that no CXR or antibiotics are necessary in routine cases (See attached algorithm). A CRP level > 100 mg/L corresponds with a substantially elevated probability of pneumonia. Thus, for patients with low and intermediate-probability of pneumonia based on clinical grounds, a CRP >100 mg/L would support CXR ordering, and for patients with high clinical suspicion, antibiotic therapy should be considered regardless of the CXR result (since studies show that CXR misses about 10% of community-acquired pneumonia confirmed with follow-up CXR or chest computed tomography). Overall, the addition of CRP test results would reduce the need for CXR ordering and antibiotic therapy in cases with an intermediate clinical probability of pneumonia and a low CRP level; and increase the need for CXR ordering and possibly antibiotic therapy in cases with intermediate or high clinical probability of pneumonia and a high CRP level. In this way, we hypothesize that the CRP-guided management algorithm will improve the proportion of patients with acute cough illness who receive appropriate diagnostic and therapeutic interventions in the ED.

We suspect that most patients with clinically apparent pneumonia will have high CRP levels. However, pneumonia can be a difficult diagnosis to make when patients present with atypical clinical manifestations (e.g. the elderly or COPD patients), or in practice settings where radiography is not readily available. In these settings, the addition of CRP testing may help identify a small number of pneumonia cases that might otherwise go undetected and result in delays in appropriate care. In the large number of patients with intermediate probability of pneumonia, such as adults with acute cough illness who have abnormal vital signs, but normal examinations, particularly in RSV and influenza season, a CRP level < 10 mg/L could provide clinically significant reassurance to refrain from further testing or empiric antibiotic treatment. A normal CRP level may also provide support to clinicians who are receiving pressure from patients to prescribe antibiotics when they are not clinically indicated. Indirect or future benefits to society are possible if research results show that CRP-guided management strategies can decrease the costs of health care.

Randomization using a random number generator will be conducted by investigators at the data coordinating center (Philadelphia, PA), and results placed in sequentially number study packets. The study personnel that enroll patients will be blinded to the randomization result until after the patient has provided informed consent to participate in the study.

Interventions

* Staff Educational Seminar: Prior to beginning the study, all staff will be informed about the performance characteristics of CRP in adults with acute cough illness, and current clinical practice recommendations regarding evaluation and treatment of acute cough illness, particularly acute bronchitis.
* CRP-Guided Algorithm: Study subjects randomized to the CRP-guided management algorithm will have a point-of-care CRP test performed shortly after triage using a finger-stick specimen. The result, along with a printed management algorithm for interpreting the CRP level (see Appendix), will be placed in the chart. The general guidelines for interpreting CRP levels will be as described above.

Human Subjects Procedures

* Recruitment and Initial Contact Method. As described above, appropriate patients will be referred to study personnel by the triage nurse. Initial contact and informed consent will be conducted in a discrete manner, and in a private setting.
* Informed consent. Will be obtained from study personnel that have been trained in Human Subjects Protection. The time involved for the research subject in obtaining informed consent is about 10 minutes.
* CRP measurement. A finger-stick blood test will be performed using the NycoCard II Reader (Axis-Shield, Norway). See testing instrument description in Appendix. The US FDA has approved the diagnostic test kit as one of moderate complexity for these specific circumstances. The CRP test will not be billed to the patient. The time involved for the research subject in performing the CRP test is about 10 minutes.
* Chart abstraction. The Chart Abstraction instrument will resemble that used in the baseline periods (11/03-2/04 and 11/04-2/05) of the currently IRB-approved study with the following modification, except that we will also abstract findings from the physical examination portion of the medical record relating to the chest examination.
* Telephone follow-up survey. Study subjects will be contacted by telephone 2-4 weeks following their emergency department visit by trained research staff using the same telephone survey instrument used in the baseline period (already approved). The time involved for the research subject in completing the telephone survey is about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 years) seeking care for an acute respiratory illness (duration < 10 days) in which cough is a chief complaint.
* Eligible patients will be required to have at least 1 symptom of acute respiratory tract infection (fever, night sweats, rhinorrhea, sinus congestion, myalgias).

Exclusion Criteria:

* Previous (within 21 days) antibiotic treatment;
* immunodeficiency;
* cystic fibrosis;
* patient requiring immediate evaluation/management;
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Chest X-ray utilization, Antibiotic treatment, Time in emergency department, Subsequent office or emergency department visits (within 2 weeks; Subsequent hospitalization, Time-to-illness resolution

SECONDARY OUTCOMES:
Satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Gonzales, MD, Principal Investigator — University of California, San Francisco; Joshua Metlay, MD, Principal Investigator — VAMC Pittsburgh
Locations (2):
- United States (2):
  - Truman Medical Center, Kansas City, Missouri
  - Veterans Affairs Medical Center, Kansas City, Missouri

REFERENCES:
- [Derived] Smedemark SA, Aabenhus R, Llor C, Fournaise A, Olsen O, Jorgensen KJ. Biomarkers as point-of-care tests to guide prescription of antibiotics in people with acute respiratory infections in primary care. Cochrane Database Syst Rev. 2022 Oct 17;10(10):CD010130. doi: 10.1002/14651858.CD010130.pub3. PMID 36250577